CLINICAL TRIAL: NCT01383785
Title: Phase 4 Study of Primary Angioplasty Combined Distal Injection of Abciximab to Thrombus and Aspiration With Catheter
Brief Title: Thrombus Aspiration for OcLuded Coronary Artery Enhanced With Distal Injection Of Abciximab
Acronym: TOLEDO1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, J.Moreu, Director catheterization laboratory, Hospital Virgen de la Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-2008/52
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Myocardial Infarction; Occlusive Thrombus
Keywords: Primary PTCA; Thrombus Aspiration Catheter; Intracoronary Abciximab
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GROUP A (Active Comparator): Intracoronary full bolus dose of abciximab proximal to thrombus occlusion
  Interventions: Other: Intracoronary direct injection
- GROUP B (Experimental): Half bolus of intracoronary abciximab proximal to thrombus occlusion and the other half distal by aspiration catheter
  Interventions: Other: Intracoronary and distal injection by aspiration device
- GROUP C (Experimental): Distal injection to thrombus occlusion of total bolus dose of abciximab by aspiration catheter
  Interventions: Other: Intracoronary distal injection by aspiration catheter device

INTERVENTIONS:
Other: Intracoronary direct injection — Abciximab bolus dosage: 0,125 mg/kg.
  Group A: Intracoronary full bolus dose of abciximab proximal to thrombus occlusion. The investigators inject the bolus of abciximab by catheter guide before cross the occlusion. This in the normal way in study' laboratory.
  Other Names: Abciximab, thrombus aspiration catheter
  Arms: GROUP A
Other: Intracoronary and distal injection by aspiration device — Abciximab bolus dosage: 0,125 mg/kg.
  Group B: Half bolus of intracoronary abciximab proximal to thrombus occlusion and the other half distal by aspiration catheter. The investigators inject half of the dose like group A and the other half like group C.
  Other Names: Abciximab, thrombus aspiration catheter
  Arms: GROUP B
Other: Intracoronary distal injection by aspiration catheter device — Abciximab bolus dosage: 0,125 mg/kg.
  Group C: Distal injection to thrombus occlusion of total bolus dose of abciximab by aspiration catheter. The investigators inject the bolus after cross the occlusion using an aspiration catheter.
  Other Names: Abciximab, thrombus aspiration catheter
  Arms: GROUP C

SUMMARY:
Aims: (to prove that) The distal injection of IIb IIIa platelet receptor blocker to the thrombus occlusion is better than normal injection during primary percutaneous intervention (PCI) for the treatment of acute myocardial infarction. Using this modification of injection method the investigators can achieve less microvascular damage and a reduction of the infarct size with a significant improvement of the outcome at six months.

DETAILED DESCRIPTION:
There are some evidence about the utilization of aspiration catheter (Indication class IIb with level of evidence B in European Guidelines) and intravenous abciximab (indication Class IIa an level of evidence A in European Guidelines) in primary PTCA. Direct intracoronary injection of abciximab get smaller infarct size than intravenous injection. The hypothesis of our study are that direct distal injection of abciximab by aspiration catheter will be better than proximal intracoronary injection with reduction in infarct size and microvascular damage quantified by Magnetic resonance (MR) and 6 months mortality.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction patients between 3 and 12 hours after symptoms onset

Exclusion Criteria:

* Hemodynamic instability
* TIMI flow 2 or 3
* Life expectance less than 6 months
* Contraindication to AAS, clopidogrel or abciximab
* Severe tortuosity of occluded vessel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Infarct size | Between 2 and 9 days after primary ptca
  Infarct size quantified by MR

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 6 months
  Cardiac mortality, reinfarction, new revascularization, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jose Moreu, Phd,MD, Principal Investigator — Hospital Virgen de la Salud. Toledo. Spain; Luis Rodriguez-Padial, Phd MD, Study Director — Hospital Virgen de la Salud
Locations (1):
- Hospital Virgen de la Salud, Toledo, Toledo, Spain

REFERENCES:
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Svilaas T, Vlaar PJ, van der Horst IC, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Thrombus aspiration during primary percutaneous coronary intervention. N Engl J Med. 2008 Feb 7;358(6):557-67. doi: 10.1056/NEJMoa0706416. PMID 18256391
- [Background] Vetrovec GW. Improving reperfusion in patients with myocardial infarction. N Engl J Med. 2008 Feb 7;358(6):634-7. doi: 10.1056/NEJMe0708910. No abstract available. PMID 18256399
- [Background] Thiele H, Schindler K, Friedenberger J, Eitel I, Furnau G, Grebe E, Erbs S, Linke A, Mobius-Winkler S, Kivelitz D, Schuler G. Intracoronary compared with intravenous bolus abciximab application in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention: the randomized Leipzig immediate percutaneous coronary intervention abciximab IV versus IC in ST-elevation myocardial infarction trial. Circulation. 2008 Jul 1;118(1):49-57. doi: 10.1161/CIRCULATIONAHA.107.747642. Epub 2008 Jun 16. PMID 18559698
- [Background] Nijveldt R, Beek AM, Hirsch A, Stoel MG, Hofman MB, Umans VA, Algra PR, Twisk JW, van Rossum AC. Functional recovery after acute myocardial infarction: comparison between angiography, electrocardiography, and cardiovascular magnetic resonance measures of microvascular injury. J Am Coll Cardiol. 2008 Jul 15;52(3):181-9. doi: 10.1016/j.jacc.2008.04.006. PMID 18617066